CLINICAL TRIAL: NCT02391376
Title: Heat Transfer by Three Types of Packs and Its Implication on the Flexibility of the Lower Back: a Randomized, Controlled Trial
Brief Title: Heat Transfer by Three Types of Packs and Its Implication on the Flexibility of the Lower Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca Nassr, PT; MSc., Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TUCM/1261/B326e/2013
Record Dates: First submitted 2015-03-03; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Physical Therapy Techniques
Keywords: superficial heat; hot pack; thermotherapy; physiotherapy; Schober Test
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- moist heat pack group (Experimental): Three sessions of 15 minutes of superficial heat through a moist heat pack on the lower back of healthy subjects
  Interventions: Other: moist heat pack; ;
- seed pack group (Experimental): Three sessions of 15 minutes of superficial heat through a seed pack on the lower back of healthy subjects
  Interventions: Other: seed pack
- gel pack group (Experimental): Three sessions of 15 minutes of superficial heat through a gel pack on the lower back of healthy subjects
  Interventions: Other: gel pack

INTERVENTIONS:
Other: moist heat pack; ; — Three sessions of 15 minutes of superficial heat through a moist heat pack-MHP applied on the lower back.
  Arms: moist heat pack group
Other: seed pack — Three sessions of 15 minutes of superficial heat through a seed pack-SP applied on the lower back.
  Arms: seed pack group
Other: gel pack — Three sessions of 15 minutes of superficial heat through a gel pack-GP applied on the lower back.
  Arms: gel pack group

SUMMARY:
The purpose of this study is to compare the effects generated by the application of three different packs on the flexibility of the lower back of sedentary students. Method: Three sessions of 15 minutes of superficial heat through a hot pack (moist heat pack-MHP, seed pack-SP or gel pack-GP) were applied on the lower back. Pack and lower back temperatures and erythema were registered every 5 minutes. Schober test was performed before first session and after the third session.

DETAILED DESCRIPTION:
A different type of hot pack was applied in the lower back of each subject: moist heat pack (MHP) , seed pack (SP) or gel pack (GP) as directed by each manufacturer and in accordance with clinical practice for 15 minutes for 3 consecutive days. On day one, prior to the application of the pack, the initial evaluation of flexibility of the lumbar spine of each subject was recorded using Schober test. On day 3, after the application of each pack, the final evaluation of the flexibility of the lower back was performed using the same test. During the sessions, the temperature of the corporal area, the temperature of the pack and the pigmentation change of the corporal area were assessed every 5 minutes through a photographic record.The method used to assess the flexibility was the Schober Test. In order to perform the evaluation, the patient was placed in standing position with its bare feet slightly apart; two points were marked on the skin, one above the spinous apophysis S1 and another point, 10 cm above that mark. The patient performed a maximal trunk flexion without flexing the knees and the increase of the distance between the two marks was recorded. After this evaluation, the packs were applied on the lower back, wrapped in two layers of towels in order to avoid skin injuries by the heat. The temperature of the lower back and of each type of pack was recorded at minutes 0 (baseline measurement), 5, 10 and 15. Temperature was measured through a digital pyrometer at a set distance of 50 cm and it was held perpendicular to patient skin and the pack. The photographic record of the lower back of each subject, before and after each session of superficial thermotherapy, was recorded using a digital camera . The camera was placed perpendicular to the lower back, at a distance of 50 cm. The brightness of the photograph was taken into account so as not to affect the later analysis of the erythema. The erythema analysis of the lower back was performed with the freeware Picture Color Analyzer (Shizuoka, Japan; http://www.isao.com). The software measures the red color intensity of each pixel (attributing a value between 1 and 255) within the chosen area. The average red color value obtained in arbitrary units is the result of the following formula: Average red color = total red color value / (255 X number of pixels in the area).

ELIGIBILITY:
Inclusion Criteria:

* sedentary subjects (physical activity performed less than 3 times-week)

Exclusion Criteria:

* recent scars or wounds in the lower back region,
* history of peripheral vascular diseases,
* impaired sensitivity,
* body mass index above 25 kg/m2,
* fat index above 14% according to Faulkner's formula.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change of lower back flexibility (Schober test) | Before first session (day 1) and after the third session (day 3-final day).
  Schober test

SECONDARY OUTCOMES:
Change of pack and lower back temperatures | every 5 minutes during each one of the three 15 minutes sessions
Change of lower back erythema | every 5 minutes during each one of the three 15 minutes sessions